CLINICAL TRIAL: NCT07042165
Title: Treatment of Bile Acid Diarrhoea With Atorvastatin (BASTA): A Randomised, Double-Blind, Placebo-Controlled, Crossover, Investigator-Initiated Trial
Brief Title: Treatment of Bile Acid Diarrhoea With Atorvastatin
Acronym: BASTA
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Asger Lund, MD (Other)
Collaborators: Fonden til Lægevidenskabens Fremme (Other); Prosektor Axel Søeborg Ohlsens Mindelegat (Other); Læge Sofus Carl Emil Friis og Hustru Olga Doris Friis' Legat (Other); Aase and Ejnar Danielsens Foundation (Other)
Responsible Party: Sponsor-Investigator, Asger Lund, MD, MD, PhD, University Hospital, Gentofte, Copenhagen
Organization: University Hospital, Gentofte, Copenhagen (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: EU trial no. 2025-521856-47-00
Record Dates: First submitted 2025-06-05; First posted 2025-06-27 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Bile Acid Diarrhea; Bile Acid Malabsorption
Keywords: Bile Acid Diarrhea; Bile Acid Malabsorption; Atorvastatin; Randomised; Placebo; 7-alpha-C4; Crossover; Double-blind; Investigator-initiated; Proof of concept
MeSH Terms: interventions — Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo tablets are manufactored by the Central Pharmacy of the Capital Region of Denmark and are identical to the IMP except with the active ingredient (atorvastatin) omitted. Participants will be administering one tablet for two weeks followed by two tablets for two weeks. Then four weeks of washout before entering the atorvastatin arm (crossover).
  Interventions: Drug: Placebo
- Atorvastatin (Experimental): 40 mg Atorvastatin tablets are manufactored by the Central Pharmacy of the Capital Region of Denmark and are identical to the placebo tablets except containing the active ingredient (atorvastatin). Participants will be administering one tablet for two weeks followed by two tablets for two weeks (80 mg atorvastatin). Then four weeks of washout before entering the placebo arm (crossover).
  Interventions: Drug: Atorvastatin

INTERVENTIONS:
Drug: Atorvastatin — Participants will be orally administering one tablet daily of 40 mg Atorvastatin for two weeks followed by two tablets daily for two weeks (totalling 80 mg daily).
  Arms: Atorvastatin
Drug: Placebo — Placebo tablets are manufactored by the Central Pharmacy of the Capital Region of Denmark and are identical to the IMP except with the active ingredient (atorvastatin) omitted. Participants will be orally administering one tablet daily for two weeks followed by two tablets daily for two weeks.
  Arms: Placebo

SUMMARY:
Bile acid diarrhoea (BAD) is a socially debilitating disease with stomach pain, high stool frequency, urgency, and faecal incontinence as the main symptoms. Studies estimate that 1-2% of the population suffers from the disease.

There is an unmet need for more treatment options in patients suffering from BAD.

The investigators hypothesise that atorvastatin treatment lowers bile acid synthesis in patients with bile acid diarrhoea. The investigators will investigate this hypothesis in the current study, BASTA, which is a Randomised, Double-Blind, Placebo-Controlled, Crossover, Proof of Concept, Investigator-Initiated, Trial.

DETAILED DESCRIPTION:
Bile acid diarrhoea (BAD) is a socially debilitating disease with stomach pain, high stool frequency, urgency, and faecal incontinence as the main symptoms. Studies estimate that 1-2% of the population suffers from the disease.

Bile acids are synthesised from cholesterol in hepatocytes through a tightly regulated enzymatic process and then excreted to the gut lumen in response to food ingestion. In a healthy individual 95 % of the bile acids are recycled in the enterohepatic circulation in a tightly regulated process. BAD symptoms arise due to a pathological spill-over of bile acids to the colon.

Currently, individuals with BAD are typically treated with bile acids sequestrants. However, only about 2/3 patients experience an improvement in their symptoms on this treatment. Thus, the possibility of yet another tool in the toolbox is compelling.

Statins are used by millions of patients world-wide to reduce their risk of cardiovascular morbidity and mortality and are considered safe with overall mild and benign adverse effects. Statins lower the intracellular levels of cholesterol in hepatocytes. As such, atorvastatin could potentially reduce the bile acid production in individuals with BAD leading to a reduction or normalisation of the amount of bile acids secreted to the intestinal lumen and entering the colon. Unpublished results from the investigators' group show a 43 % reduction of serum C4, a biomarker of bile acid synthesis which can also be used to diagnose BAD, in healthy, young men, who were treated with atorvastatin for 14 days (7 days of 40 mg atorvastatin once daily followed by 7 days of 80 mg atorvastatin once daily) compared to placebo treatment.

The investigators hypothesise that atorvastatin treatment lowers bile acid synthesis in patients with bile acid diarrhoea.

The current study aims to investigate whether atorvastatin treatment lowers the synthesis of bile acids, measured via the well-known bile acid synthesis marker C4, in a dose-response manner in patients with severe bile acid diarrhoea. The investigators expect the reduction of bile acid synthesis to lead to a reduction in bile acid diarrhoea symptoms since the pathophysiology of the disease is a spill-over of bile acids to the colon. Specifically, the primary endpoint is the reduction in percentage of C4 at the end of the 80 mg treatment period compared to placebo. Additionally, the investigators will investigate the effect of atorvastatin treatment in patients with severe bile acid diarrhoea on symptoms, hepatobiliary markers, metabolic markers, glycaemic control markers, stool samples and safety.

ELIGIBILITY:
Inclusion Criteria:

* age 18 years or above
* Self-identification as White
* Confirmed moderate-severe bile acid diarrhoea with a SeHCAT test result of ≤ 10 %
* Reported number of average daily stools ≥ 3 stools per day
* Reported number of average daily watery (6 or 7 on the Bristol Stool Chart) stools ≥ 1 stools per day(30)
* Informed and written consent

Exclusion Criteria:

* Unwillingness to pause any of the following medications during the trial: bile acid sequestrants, morphine medication, liraglutide or anti-constipation medication (e.g., lactulose, laxoberal, magnesia)
* Unwillingness to pause any anti-diarrhoea medication (e.g., imodium) from 3 days before initiation of each stool diary until after the respective visit
* If regularly administering psyllium or metformin, unwillingness to agree to a stable dose of psyllium or metformin throughout the trial
* Concomitant use of any drug in the GLP-1 receptor agonist drug class with the exception of paused liraglutide, see above
* Concomitant use of any kind of insulin medication
* Planned major changes in food consumption throughout the trial, including planned weight loss attempts
* Prior use of any statin within the recent 6 months
* Intake of larger quantities of grapefruit juice during trial participation, at the discretion of the investigator
* History of/present hepatobiliary disorder (except for simple metabolic dysfunction-associated fatty liver disease) and/or alanine aminotransferase and/or serum aspartate aminotransferase ≥ 3 times upper limit of normal
* Crohn's disease, ulcerative colitis, celiac disease or lactose intolerance
* Previous intestinal resection or major intra-abdominal surgery incl. stoma (cholecystectomy and appendectomy not included)
* Nephropathy with estimated glomerular filtration rate < 45 ml/min/1,73 m2
* Plasma level of creatine kinase ≥ 5 times the upper limit of normal
* A recent stroke or transient ischemic attack (within 6 months)
* Any treatment or condition requiring acute or subacute medical or surgical intervention
* Hypothyroidism or hyperthyroidism, if not well regulated, at the discretion of the investigator
* Active or recent (within 6 months) clinically significant malignant disease (non-melanoma skin cancer not included), at the discretion of the investigator
* Alcohol consumption exceeding 12 units/week for women or 18 units/week for men, respectively. These thresholds are based on the limits of the European Association for the Study of the Liver
* Drug abuse, at the discretion of the investigator
* Fertile women not using any of the following contraceptive methods for the duration of the trial until at least 5 days after end of trial: Hormonal (tablet/pill, depot injection of progesterone, subdermal gestagen implantation, hormone intrauterine devices (IUD), hormonal vaginal ring or transdermal hormonal patch) associated with inhibition of ovulation, chemical (copper IUD), sterilisation, vasectomised partner with a confirmatory test, or sexual abstinence per the investigator's discretion
* Pregnant or nursing women
* Known or suspected hypersensitivity to atorvastatin or any of the additives in the tablet
* Receipt of any investigational drug within 30 days prior to visit 0
* Concomitant treatment with any of the following (topical administration not included): ciclosporin, telithromycin, clarithromycin, delavirdin, stiripentol, ketoconazol, voriconazol, itraconazol, posaconazol, letermovir, ritonavir, lopinavir, atazanavir, indinavir, darunavir, bocepravir, telaprevir, elbasvir/grazoprevir, ledipasvir/sofosbuvir, erythromycin, niacin, ezetimibe, fusidic acid, gemfibrozil, colchicine, digoxin, warfarin
* Unable to speak or understand Danish or mental incapacity that preclude adequate understanding or cooperation or unwillingness to comply with trial requirements
* Active participation in any other clinical intervention trial (observational studies not included)
* Other concomitant disease or treatment that according to the investigator's assessment makes the person unsuitable for study participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-10-15 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Reduction in bile acid synthesis measured via 7alpha-Hydroxy-4-cholesten-3-on (C4) | The end of week 4 and the end of week 12.
  Ratio of geometric mean concentration of 7alpha-Hydroxy-4-cholesten-3-on (C4) at the end of the 80 mg atorvastatin treatment period compared to the end of the placebo treatment period.

SECONDARY OUTCOMES:
Reduction in bile acid synthesis measured via C4 | The end of week 4 and the end of week 12.
  Difference in mean concentration of 7alpha-Hydroxy-4-cholesten-3-on (C4) in μg/L at the end of the 80 mg atorvastatin treatment period compared to the end of the placebo treatment period.
Reduction in BAD symptoms measured via a stool diary. | Week 4 and week 12.
  Difference in mean daily stools during the last week of the 80 mg atorvastatin treatment period compared to the last week of the placebo treatment period as assessed by a 7-day stool diary
A reduction in BAD symptoms measured via a stool diary. | Week 4 and week 12.
  Difference in mean daily watery stools during the last week of the 80 mg atorvastatin treatment period compared to the last week of the placebo treatment period as assessed by the total watery (6 or 7 on the Bristol Stool Chart) stools in a 7-day stool diary
Symptom severity measured via IBS-SSS | The end of week 4 and the end of week 12.
  Difference in symptom severity measured via a danish translation of the validated questionnaire Irritable Bowel Syndrome Symptom Severity Score (IBS-SSS).
  The answers are on a scale of 0-500, where a higher score indicates worse symptoms.
Reduction in bile acid synthesis measured via C4. | The end of week 4 and the end of week 12.
  Proportion of patients with a reduction of 7alpha-Hydroxy-4-cholesten-3-on (C4) below 31 μg/L (%)
Reduction in bile acid synthesis measured via C4 | The end of week 4 and the end of week 12.
  Proportion of patients with a reduction of 7alpha-Hydroxy-4-cholesten-3-on (C4) below 46 μg/L (%)
Bile acid metabolism measured via FGF-19 | The end of week 4 and the end of week 12.
  Fibroblast growth factor 19 (FGF-19) (pg/mL)
Bile acid metabolism measured via blood levels of total bile acids | The end of week 4 and the end of week 12.
  Blood levels of total bile acids (μmol/L)
Cholesterol metabolism | The end of week 4 and the end of week 12.
  Total cholesterol (mmol/L)
Cholesterol metabolism | The end of week 4 and the end of week 12.
  Low-density lipoprotein (LDL) cholesterol (mmol/L)
Bile acid levels measured in stool samples | The end of week 4 and the end of week 12.
  Stool sample levels of total bile acids (μmol/g)

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Clinical Metabolic Research, Gentofte Hospital, Hellerup, Denmark

IPD SHARING:
Plan to Share IPD: Undecided